CLINICAL TRIAL: NCT04257851
Title: Is Theophylline More Effective Than Sumatriptan in the Treatment of Post-dural Puncture Headache: A Randomized Clinical Trial
Brief Title: Is Theophylline More Effective Than Sumatriptan in the Treatment of Post-dural Puncture Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DTH: 20001
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2020-02

CONDITIONS: Post-Dural Puncture Headache
Keywords: Post-dural puncture headache; Spinal anesthesia; Sumatriptan; Theophylline
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Theophylline; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (n=30) (Active Comparator): Theophylline group
  Interventions: Drug: Theophylline Anhydrous Oral Tablet
- Group S (n=30) (Active Comparator): Sumatriptan group
  Interventions: Drug: Sumatriptan Succinate Oral Tablet

INTERVENTIONS:
Drug: Theophylline Anhydrous Oral Tablet — Theophylline tablet (150 mg/12h)
  Other Names: Quibron-T/SR tablets
  Arms: Group T (n=30)
Drug: Sumatriptan Succinate Oral Tablet — Sumatriptan tablet (25 mg/12h)
  Other Names: Sumigran tablets
  Arms: Group S (n=30)

SUMMARY:
Objectives: To compare the safety and efficacy of oral theophylline versus oral sumatriptan in the treatment of post-dural puncture headache (PDPH).

Background: PDPH is the most frequent complication of procedures associated with dural puncture for spinal anesthesia or following accidental dural puncture during epidural anesthesia. Since invasive treatments have known complications, pharmacologic management may be preferable.

Patients and Methods: This was a prospective, randomized, double-blind, phase four clinical trial; carried out on 60 patients presented with PDPH at our hospital. Patients were randomly allocated into two equal groups (30 patients each); group T, received oral theophylline, and group S, received oral sumatriptan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NPRS score of ≥ 5
* American Society of Anesthesiologists (ASA) physical status ≤ II
* Age from 21 to 50 years

Exclusion Criteria:

* Patients with NPRS score < 5
* ASA physical status > II
* Age < 21 years or > 50 years
* Pregnant women
* History of; Chronic headache, Cluster headache, Migraine
* History of; Convulsions, Cerebrovascular accident, Previous neurological diseases
* History of peripheral vascular disease (ischemic colitis)
* Signs of meningismus
* Dysrhythmia
* Hypertension
* Ischemic heart disease
* Hyperthyroidism
* Liver or Renal impairment
* Use of selective serotonin reuptake inhibitors (SSRIs)
* Use of ergotamine derivatives in the past 24 hours
* Use of monoamine oxidase inhibitors (MAOIs) in the last two weeks
* Use of any kind of opiates
* Allergy to the study medications
* Any contraindication of oral intake

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Median and Range of Numeric Pain Rating Scale (NPRS) score [(median (range)] | 48 hours after initiation of treatment
  NPRS measures the severity of PDPH, it is a 11 point scale from 0-10; where 0=No pain and 10=Worst possible pain (before, 2h, 6h, 12h, 18h, 24h, then every 12h till 48h)
Mean and Standard deviation of Numeric Pain Rating Scale (NPRS) score (mean±SD) | 48 hours after initiation of treatment
  NPRS measures the severity of PDPH, it is a 11 point scale from 0-10; where 0=No pain and 10=Worst possible pain (before, 2h, 6h, 12h, 18h, 24h, then every 12h till 48h)

SECONDARY OUTCOMES:
Mean and Standard deviation of PDPH duration (hours) (mean±SD) | 48 hours after initiation of treatment
  Time from PDPH onset till NPRS score ≤ 3
Mean and Standard deviation of Length of hospital stay (days) (mean±SD) | 48 hours after initiation of treatment
  Time from hospital admission till discharge
Number of participants and Rate of Treatment-related side effects | 48 hours after initiation of treatment
  Number of participants and Rate of: Palpitation, Dizziness, Gastric irritation, Nausea/Vomiting, Diarrhea, Warm sensations in the body, Tingling sensation, and Tightness in the chest, throat, neck, or jaws.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt